CLINICAL TRIAL: NCT01748188
Title: Valuation of the Dexketoprofen Effectiveness on Subacromial Syndrome With Different Physiotherapy Treatments.
Brief Title: The Effectiveness of Dexketoprofen on Shoulder Pain Using Different Physiotherapy Treatments
Acronym: DOFIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Principal Investigator, Rosa Sola, University Professor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URV
Record Dates: First submitted 2012-10-28; First posted 2012-12-12 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Shoulder Pain
Keywords: Subacromial syndrome; Dexketoprofen; Phonophoresis; Iontophoresis; Ultrasounds; VAS; DASH score; Constant score
MeSH Terms: conditions — Shoulder Pain | interventions — High-Energy Shock Waves; Phonophoresis; Iontophoresis; Exercise; Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ultrasound + Exercises + Cryotherapy (Active Comparator): Ultrasound of 1 Megahertz (MHz), intensity 2 W/cm2, 5 minutes, for 20 sessions.
  Interventions: Procedure: Ultrasound; Procedure: Exercises; Procedure: Cryotherapy
- Phonophoresis + Exercises + Cryotherapy (Experimental): Phonophoresis with 50 mg dexketoprofen (Enangel), 1 MHz, intensity 2 W/cm2, 5 minutes, for 20 sessions.
  Interventions: Procedure: Phonophoresis; Procedure: Exercises; Procedure: Cryotherapy
- Iontophoresis + Exercices + Cryotherapy (Experimental): Iontophoresis by galvanic direct current with 50 mg dexketoprofen (Enantyum), intensity 2 milliamperes (mA), 20 minutes, for 20 sessions.
  Interventions: Procedure: Iontophoresis; Procedure: Exercises; Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound of 1 MHz, intensity 2 W/cm2, 5 minutes, for 20 sessions.
  Arms: Ultrasound + Exercises + Cryotherapy
Procedure: Phonophoresis — Phonophoresis with 50 mg dexketoprofen (Enangel), 1 MHz, intensity 2 W/cm2, 5 minutes, for 20 sessions.
  Arms: Phonophoresis + Exercises + Cryotherapy
Procedure: Iontophoresis — Iontophoresis by galvanic direct current with 50 mg dexketoprofen (Enantyum), intensity 2 mA, 20 minutes, for 20 sessions.
  Arms: Iontophoresis + Exercices + Cryotherapy
Procedure: Exercises — Guideline of 7 standardized exercises to improve the muscular force and to open the subacromial space.
Procedure: Cryotherapy — Cooling located by a cold air bundle to -32 Celsius degrees (ºC) for 3 minutes.

SUMMARY:
The purpose of this study is to determine whether dexketoprofen administered by phonophoresis or iontophoresis is more effective in the treatment of subacromial syndrome that the conventional therapy with ultrasounds.

DETAILED DESCRIPTION:
It is a question of valuing the decrease of the pain (by means of the visual analogic scale pain score) and the increase of the functionality of the joint (by means of Dash and Constant scores) of three different treatments from physical therapy to establish the most effective protocol for the treatment of the subacromial syndrome.

Determine the best physiotherapy treatment for subacromial syndrome with 20 sessions of different treatments.

A group will receive the conventional treatment with ultrasounds without drugs, another group will receive dexketoprofen by phonophoresis and the third group will receive dexketoprofen by iontophoresis.

ELIGIBILITY:
Inclusion Criteria:

* Subacromial syndrome diagnosed by ultrasound scanning with Rotator cuff tendinitis or partial break of the rotator cuff and / or of the brachial biceps.
* Informed consent.

Exclusion Criteria:

* To suffer shoulder arthritis or any shoulder pathology with mobility limitation.
* Fibromyalgia
* Psychologic or psychiatric pathologies
* Hypersensibility to the drug
* Back or shoulder traumatism
* To have received an analgesic infiltration on the affected shoulder in the last month
* Lack of adherence to the treatment upper to 15 % of the sessions

Ages: 36 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pain measure by the visual analogic scale pain score. | 1 month

SECONDARY OUTCOMES:
Functionality of the joint by Dash and Constant scores | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Carme Casajuana, PT, Study Director — Hospital Universitari Sant Joan de Reus
Locations (1):
- Hospital Universitari Sant Joan, Reus, Tarragona, Spain

REFERENCES:
- [Derived] Perez-Merino L, Casajuana MC, Bernal G, Faba J, Astilleros AE, Gonzalez R, Giralt M, Romeu M, Nogues MR. Evaluation of the effectiveness of three physiotherapeutic treatments for subacromial impingement syndrome: a randomised clinical trial. Physiotherapy. 2016 Mar;102(1):57-63. doi: 10.1016/j.physio.2015.01.010. Epub 2015 Mar 25. PMID 26051846